CLINICAL TRIAL: NCT02073617
Title: Aortic Valve and Root Measurements Under Real-Time 3-Dimensional Visualization During Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-00804
Record Dates: First submitted 2014-02-19; First posted 2014-02-27 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Coronary Artery Disease; Aortic Stenosis
Keywords: DynaCT; Aortic valve and root measurements; TAVR
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Real-time 3-dimensional DynaCT (Experimental): Patients will undergo the standard CTA protocol and invasive coronary angiography performed as part of the pre-operative assessment for TAVR. Patients in this study will also undergo DynaCT during coronary angiography, utilizing 1 acquisition sweep and 20 to 35cc more of contrast media. Measurements of the major aortic annulus diameter, orthogonal minor aortic annulus diameter, aortic annulus perimeter, maximum ascending aorta diameter at 40mm above the annulus, sinus of Valsalva diameters, sinus of Valsalva heights, and aortic root angulation will be made using both the CTA and DynaCT protocols by a radiologist blinded to patient identity. Based on these measurements, a trained interventional cardiologist will select the appropriate TAVR size for the patient.
  Interventions: Radiation: Real-time 3-dimensional DynaCT

INTERVENTIONS:
Radiation: Real-time 3-dimensional DynaCT — After coronary angiography is performed, a 6Fr pigtail catheter will be placed in the aorta and 40cc of 50% contrast media diluted normal saline will be delivered using standard automated injection during dynaCT cardiac image acquisition. Intravenous delivery of contrast as alternative.

SUMMARY:
The American College of Cardiology/American Heart Association guidelines place symptomatic severe Aortic Stenosis as a class I indication for aortic valve replacement. With the recently approved Edwards-Sapien TAVR device and the ongoing investigations using the CoreValve TAVR device, patients ineligible or at high risk for open-heart surgery are now eligible to undergo TAVR.

Patients selected for TAVR undergo an EKG-gated cardiac Multislice CTA to evaluate aortic valve anatomy and aortic root dimensions for device sizing, as well as coronary angiography to define coronary anatomy. Both tests utilize contrast media to visualize anatomy, which may result in contrast-induced nephropathy in anywhere from 7.5% to more than 50% of patients depending on associated clinical risk factors.

There is a need to consolidate this pre-operative testing whenever possible, and with real-time 3-dimensional visualization of aortic valve and root anatomy using DynaCT cardiac acquisition in the cath lab angiography suite during the coronary angiography, there may be a benefit with reduced contrast load (20 to 35cc for DynaCT, 100cc for CTA).

We would like to make a comparison of aortic valve and root measurements using CTA and DynaCT to affirm the accuracy of DynaCT vs the CTA gold standard.

DETAILED DESCRIPTION:
Calcific or degenerative aortic valve disease is one of the most common valvular diseases among the elderly and, with life expectancy continuing to increase, a major source of burden on current healthcare. Although patients with aortic stenosis (AS) can remain asymptomatic for a prolonged period, they do eventually develop symptoms, including angina, exertional syncope and heart failure, which is associated with a 5-year, 3-year, and 1-year, respectively, 50% mortality. The American College of Cardiology/American Heart Association guidelines place symptomatic severe AS as a class I indication for aortic valve replacement. Currently, surgical replacement of the aortic valve is the standard of care. However, with the recently approved Edwards-Sapient TAVR device and the ongoing investigations using the CoreValve TAVR device, patients ineligible or at high risk for open-heart surgery are now eligible to undergo TAVR.

Currently, patients selected for TAVR undergo an EKG-gated cardiac Multislice CTA to evaluate aortic valve anatomy and aortic root dimensions for device sizing. Patients also undergo coronary angiography to define coronary anatomy. Both tests utilize contrast media to visualize anatomy, which may result in contrast-induced nephropathy in anywhere from 7.5% to more than 50% of patients depending on associated clinical risk factors. Contrast-induced nephropathy can, in turn, lead to dialysis and/or increased mortality.

There is a need to consolidate this pre-operative testing whenever possible, and with real-time 3-dimensional visualization of aortic valve and root anatomy using DynaCT cardiac acquisition in the cath lab angiography suite during the coronary angiography, there may be a benefit with reduced contrast load (20 to 35cc for DynaCT, 100cc for CTA). DynaCT conducts fully automatic aortic root segmentation and overlays 3-dimensional structures onto 2-dimensional fluoroscopy in a few seconds (~5 seconds, 60 frames/second rotational angiography). The software automatically recognizes and represents the aortic root, detects and indicates coronary ostia and lowest cusp points of aortic valve (nadir points), and reconstructs commissure lines of aortic valve. Due to cardiac motion, 3-dimensional images without motion correction or cardiac gating will look blurred. Therefore, DynaCT reconstruction motion correction software will be used. The DynaCT motion correction software is a new algorithm that will correct for this motion and apply it during reconstruction- allowing the user to spin without using rapid pacing. However, first, a comparison of aortic valve and root measurements using CTA and DynaCT must be made to affirm the accuracy of DynaCT vs the CTA gold standard.

Study Design This is a pilot study evaluating patients undergoing TAVR at the New York University (NYU) Langone Medical Center. Patients will undergo the standard CTA protocol and invasive coronary angiography performed as part of the pre-operative assessment for TAVR. However, patients in this study will also undergo DynaCT during coronary angiography, utilizing 1 acquisition sweep and 20 to 35cc more of contrast media. Measurements of the major aortic annulus diameter, orthogonal minor aortic annulus diameter, aortic annulus perimeter, maximum ascending aorta diameter at 40mm above the annulus, sinus of Valsalva diameters, sinus of Valsalva heights, and aortic root angulation will be made using both the CTA and DynaCT protocols by a radiologist blinded to patient identity after the study has reached its target recruitment. Based on these measurements, a trained interventional cardiologist will select the appropriate TAVR size in a similarly blinded fashion after the study has reached its target recruitment (i.e. the data collected using DynaCT will not be used in the clinical decision making process). Data will be compared from both modalities using appropriate tests of reproducibility and correlation.

Study Technique CTA will be performed per standard methods as part of standard pre-TAVR evaluation.

Coronary angiography will be performed via femoral artery access (minimum 6Fr) as per standard pre-TAVR evaluation. After coronary angiography is performed, a 6Fr pigtail catheter will be placed in the aorta and 40cc of 50% contrast media diluted normal saline will be delivered using standard automated injection during dynaCT cardiac image acquisition. Intravenous delivery of contrast was considered as alternative.

As per standard care, intravenous access will be obtained and participants will be hydrated during the CTA, coronary angiography, and dynaCT procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be more than 18 years of age with a plan to undergo TAVR.

Exclusion Criteria:

* Subjects will be excluded if they meet one of the following criteria:

  1. estimated glomerular filtration rate <40 mL/min/1.73m2;
  2. highly irregular heart rates, frequent extra systoles, additional extra pulsations, not in sinus heart rhythm;
  3. allergy to contrast media;
  4. pregnant; or
  5. Unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Correlation of aortic annulus measurement measured on invasive 3D dyna CT (experimental) and on non-invasive CT scan (standard of care) | 1 day
  Each patient will undergo non-invasive CT scan for aortic annulus measurement (in order to choose appropriate TAVR size) as per standard of care. They will then undergo invasive dyna CT for aortic annulus measurement during their clinically-indicated invasive coronary angiogram. The primary outcome is correlation between the aortic annulus dimension measurement made on dyna CT and non-invasive CT.

SECONDARY OUTCOMES:
TAVR size | 1 day
  A trained interventional cardiologist will evaluate the measurements made from each CTA abd DynaCT image and select the appropriate TAVR size in a blinded fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Medical Center, New York, New York, United States